CLINICAL TRIAL: NCT04934631
Title: Testing the Utility of a Clinician Competence Scale for Therapists Using Evidence-based Cognitive Behavioural Therapy With Eating Disorder Patients
Brief Title: Testing the Utility of a Competence Scale for CBT-ED Therapists
Status: Withdrawn | Type: Observational
Why Stopped: Unable to recruit NHS sites
Sponsor: University of Sheffield (Other)
Responsible Party: Principal Investigator, Jessica Beard, Research Assistant, University of Sheffield
Other Study IDs: 298732
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Measurement Reliability; Clinician Competence
Keywords: CBT; CBT-ED; CBTS-ED; Competence; Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CBT-ED trainees and therapists.: Qualified clinicians delivering CBT-ED throughout a variety of treatment settings, working with adult eating disorder patients. Clinicians will audio-record CBT-ED therapy sessions with their eating disorder patients.
  Interventions: Other: Recording of CBT-ED session.
- Eating Disorder patients.: Adult (18+ years) eating disorder patients currently accessing CBT-ED from one of the CBT-ED therapists/trainees stated above. Patients will have one of their therapy sessions audio-recorded.
  Interventions: Other: Recording of CBT-ED session.
- Raters/Judges.: Either experts or non-experts in the field of CBT-ED. Raters will use the CBTS-ED to assess clinician competence when listening to the therapy session audio-recordings.
  Interventions: Other: Assessment of CBT-ED clinician competence.

INTERVENTIONS:
Other: Recording of CBT-ED session. — Therapists will deliver treatment as usual (CBT-ED) to eating disorder patients. Therapy session will be audio recorded.
  Groups: CBT-ED trainees and therapists.; Eating Disorder patients.
Other: Assessment of CBT-ED clinician competence. — Independent raters will assess CBT-ED competence using the Cognitive-Behavioural Therapy Scale for Eating Disorders (CBTS-ED).
  Groups: Raters/Judges.

SUMMARY:
This study aims to test the utility of a newly developed clinician competence scale for those delivering Cognitive-Behaviour Therapy for Eating Disorders (CBT-ED), specifically assessing the inter-rater reliability of the measure.

DETAILED DESCRIPTION:
Cognitive-behavioural therapy for eating disorders (CBT-ED) is currently one of the NICE (2017) recommended treatments for anorexia nervosa and the only treatment recommended for bulimia nervosa, binge-eating disorder and other specified feeing and eating disorders. When clinicians adhere to evidence-based CBT-ED treatment manuals, CBT-ED has shown demonstrable levels of effectiveness in a range of eating disorders, comparable to outcomes in controlled research settings. A key component of CBT-ED found so effective in the treatment of eating disorders is a stronger focus on behavioural change tasks which is key for changing biased thinking. However, clinicians often drift from using behavioural change components and instead focus more on the cognitive aspects of therapy, or indeed drift away from treatment manuals substantially. Therefore, a suitable measure that can accurately assess how well a clinician is delivering the therapeutic competences that ensures patients are receiving evidence-based CBT-ED thus providing them with the best chance of reaching maximum recovery is important. Whilst numerous scales have been developed, none have yet been found suitable for eating disorders, as they do not have a strong focus on the key behavioural aspects of CBT-ED. Therefore, a team of clinical researchers developed the Cognitive Behaviour Therapy Scale for Eating Disorders (CBTS-ED). This pilot study will use CBT-ED therapy session audio-recordings, and different expert and non-expert raters to a) assess the inter-rater reliability of the CBTS-ED and b) assess whether the CBTS-ED can accurately detect improvement in competence among clinicians currently undergoing post-graduate diploma training in CBT-ED. The findings from this study will provide information about the reliability of the CBTS-ED scale and its possible future uses in predicting patient outcomes.

National Institute for Health and Care Excellence (2017). Eating disorders: recognition and treatment (NICE guideline NG69). Available at: https://www.nice.org.uk/guidance/ng69

ELIGIBILITY:
Therapist Inclusion Criteria:

* Qualified clinicians with a core National Health Service (NHS) profession currently undergoing post-graduate diploma training in CBT-ED at either the University of Sheffield or University College London (UCL), or;
* Qualified clinicians not on the CBT-ED training course but delivering CBT-ED
* Treating adult (18+ years) eating disorder patients
* Have a good understanding of written and verbal English

Patient Inclusion Criteria:

* Primary diagnosis of an eating disorder
* Accessing CBT-ED
* Aged 18+ years
* Have a good understanding of written and verbal English
* Have the capacity to provide written informed consent

Rater Inclusion Criteria:

* Specialists in the field of CBT-ED, or;
* Qualified clinicians who do not ordinarily work with eating disorder patients, or;
* CBT-ED trainees at Sheffield University or UCL, or;
* CBT-ED training course supervisors at Sheffield University or UCL
* Have a good understanding of written and verbal English

Therapist Exclusion Criteria:

* Non-qualified clinicians
* Non CBT-ED clinicians
* Clinicians only treating children or young people with eating disorders (aged 17 years or younger)
* Have little understanding of written and verbal English

Patient Exclusion Criteria:

* Non-eating disorder patients
* Eating disorder patients who are accessing treatment other than CBT
* Aged 17 years or younger
* Have little understanding of written and verbal English
* Lack the capacity to understand the project and provide written informed consent

Rater Exclusion Criteria:

- Little understanding of written and verbal English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinicians delivering Cognitive-Behavioural Therapy for Eating Disorders (CBT-ED) will be assessed by independent raters using the Cognitive-Behavioural Therapy Scale for Eating Disorders (CBTS-ED). Clinicians will be delivering therapy in either NHS or Non-NHS organisations. A number of clinicians will be undergoing post-graduate diploma training in CBT-ED at either the University of Sheffield or UCL.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Reliability of the CBTS-ED | 12 months
  Internal reliability of the CBTS-ED (Cronbach's Alpha) and the inter-rater reliability of the CBTS-ED (weighted Kappa statistic).

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Waller, Principal Investigator — University of Sheffield